CLINICAL TRIAL: NCT03759756
Title: Application of Artificial Intelligence for Early Diagnosis of Esophageal Squamous Cell Carcinoma During Optical Enhancement Magnifying Endoscopy
Brief Title: Artificial Intelligence for Early Diagnosis of Esophageal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2018SDU-QILU-2
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Artificial Intelligence; Optical Enhancement Endoscopy; Magnifying Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AI visible group: the endoscopic novices analyzing the images can see the automatic diagnosis of AI during the process
  Interventions: Other: AI presentation
- AI invisible group: the endoscopic novice analyzing the images can not see the automatic diagnosis of AI during the process
  Interventions: Other: no AI presentation

INTERVENTIONS:
Other: AI presentation — AI presentation means the automatic diagnosis information of AI and AI presentation means it is visible in the group.
  Groups: AI visible group
Other: no AI presentation — AI presentation means the automatic diagnosis information of AI and no AI presentation means it is invisible in the group.
  Groups: AI invisible group

SUMMARY:
Esophageal squamous cell carcinoma is one of the most common malignant tumor of upper digestive tract. However, the detection rate and diagnosis accuracy of early esophageal squamous cell cancer is low. The aim of this study is to develop a computer-assisted diagnosis tool combining with optical magnifying endoscopy for early detection and accurate diagnosis of it.

ELIGIBILITY:
Inclusion Criteria:

* high risk patients for esophageal cancer aged 18 years or older;
* Histologically verified early esophageal squamous cell cancer.

Exclusion Criteria:

* patients whose images of esophagus not suitable for the training, validation and testing the computer-assist diagnosis tool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who came to Qilu Hospital of Shandong University and received optical magnifying OE endoscopy examination
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
the diagnosis efficiency of the AI model | 12 months
  the sensitivity, specificity and accuracy of the AI model

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PHD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China